CLINICAL TRIAL: NCT07092982
Title: Comparison of the Effects of Ultrasound-Guided Adductor Canal Block With iPACK (Space Between the Popliteal Artery and the Posterior Knee Capsule) Block Combination and Suprainguinal Fascia Iliaca Block on Postoperative Pain and Stress Response in Patients Undergoing Total Knee Arthroplasty
Brief Title: Comparison of Two Different Regional Anesthetic Methods in Total Knee Arthroplasty Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SB Istanbul Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Kubilay Ekinci, Anesthesiology and Reanimation Resident, SB Istanbul Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 56
Record Dates: First submitted 2025-07-18; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Total Knee Arthroplasty; Ultrasound Guided Supra-inguinal Fascia Iliaca Block; Adductor Canal Block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound Guided Fascia Iliaca Block (Active Comparator): Suprainguinal fascia iliaca block was applied to the patients in this group at the end of the operation.
  Interventions: Procedure: Ultrasound Guided Suprainguinal Fascia Iliaca Block
- Ultrasound Guided Adductor Canal Block + iPACK Block (Active Comparator): Adductor Canal Block and iPACK Block was applied to the patients in this group at the end of the operation.
  Interventions: Procedure: Ultrasound Guided Adductor Canal Block; Procedure: Ultrasound Guided iPACK Block

INTERVENTIONS:
Procedure: Ultrasound Guided Suprainguinal Fascia Iliaca Block — Ultrasound Guided Suprainguinal Fascia Iliaca Block, 30 ml Bupivacain %0,25
  Arms: Ultrasound Guided Fascia Iliaca Block
Procedure: Ultrasound Guided Adductor Canal Block — Ultrasound Guided Adductor Canal Block, 15ml Bupivacain %0,25
  Arms: Ultrasound Guided Adductor Canal Block + iPACK Block
Procedure: Ultrasound Guided iPACK Block — Ultrasound Guided iPACK Block, 15ml Bupivacain %0,25
  Arms: Ultrasound Guided Adductor Canal Block + iPACK Block

SUMMARY:
Total Knee Arthroplasty patients are among the orthopedic cases that experience severe postoperative pain. In these cases, pain must be controlled. If pain is not controlled, early mobilization cannot be achieved. This can result in delayed physical therapy, prolonged hospital stays, the development of nosocomial infections, and impaired cognitive function. All of these factors contribute to increased patient care costs. Multimodal analgesia methods are used to control this pain. One of these methods is peripheral nerve blocks. Peripheral nerve blocks provide pain control and reduce the likelihood of opioid use and related side effects such as nausea, vomiting, and constipation. Current studies recommend Adductor Canal Blocks and iPACK (space between the popliteal artery and the posterior knee capsule) blocks for Total Knee Arthroplasty patients. In addition, studies are also being conducted on the application of the Suprainguinal Fascia-Iliaca Block in Total Knee Arthroplasty patients. The differences in postoperative analgesic effects between these methods are a matter of interest. No study has been conducted comparing the effects of these two approaches, which are routinely applied in our clinic and comply with guidelines, on the postoperative stress response. Regional anesthesia provides adequate pain control and has a positive effect on the stress response. The investigators aim to see a similar effect in peripheral nerve blocks. Therefore, comparing the methods that mentioned will contribute to the literature. In this study, the effects of these two different approaches on postoperative stress response and analgesic efficacy will be compared in terms of patients' postoperative opioid consumption, pain at rest and with movement, time to first analgesic need and development of motor block. IL-6 and CRP values will be examined pre-operatively and post-operatively to measure the effects on the stress response.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total knee arthroplasty
* Patients aged 18-75
* Patients with ASA I-II-III

Exclusion Criteria:

* Coagulation disorders
* Allergy to local anesthetics
* Liver and renal failure
* Alcohol and drug addiction
* Cognitive dysfunction that may prevent pain assessment
* Systemic or needle insertion site infection
* Analgesic use for more than 3 months
* Patient refusal to participate in the study/refusal to consent
* Presence of a hematoma, hernia, neoplasm, etc. in the area where the block will be performed
* Pre-existing neurological deficit
* Patients with contraindications to nerve block

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-08-04 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Cumulative opioid consumption | 24 hours
  Tramadol consumption will be recorded for 24 hours.

SECONDARY OUTCOMES:
Numeric rating scale for pain | Up to 24 hours
  Variations in the Numeric Rating Scale (NRS) scores, both at rest and during movement, will be documented at specific time points (End of the surgery, Post-operative 6th, 12th and 24th hour). The NRS is a simple, single-dimensional tool used to assess pain intensity in adult patients. It is a numeric adaptation of the Visual Analog Scale (VAS), where individuals are asked to choose an integer between 0 and 10 that best represents their pain level. A score of '0' corresponds to "no pain," while '10' indicates the "worst imaginable pain" or "pain as severe as possible.
Time to first postoperative analgesic requirement | Up to 24 hours
  The time to first postoperative analgesic requirement was recorded.
Postoperative quadriceps muscle strength | Up to 24 hours
  Muscle strength assessment will be performed using the Modified Bromage Scale. (End of the surgery, Post-operative 6th, 12th and 24th hour) Grade 0: No motor block; the patient is able to fully flex the hip and knee. Grade 1: Partial motor block; the patient is able to move the knee and foot but is unable to lift the extended leg.
  Grade 2: Nearly complete motor block; the patient is unable to flex the knee and can only move the foot.
  Grade 3: Complete motor block; the patient is unable to move the ankle or the great toe.
Incidence of postoperative nausea and vomiting | Up to 24 hours
  Opioid side effects were recorded.
Quality of Recovery 15 (QoR-15) | 24 hours
  The influence of surgical and anesthetic interventions on perioperative quality of life and the patient's ability to return to routine daily activities will be systematically evaluated.
  QoR-15 has 15 questions. Each question is answered on a scale of 1 to 10. A higher score indicates more positive outcomes.
Inflammatory marker levels | Up to 24 hours
  The levels of inflammatory biomarkers (interleukin-6, CRP, NLR [Neutrophil-Lymphocyte Ratio], PLR [Platelet-Lymphocyte Ratio]) will be assessed prior to surgery and at 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- SB Istanbul Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Beginning 6 months and ending 3 years after the publication of results

REFERENCES:
- See also: Related Info — https://journals.lww.com/anesthesia-analgesia/abstract/2019/08000/addition_of_infiltration_between_the_popliteal.36.aspx